CLINICAL TRIAL: NCT03620578
Title: A Phase II Study Evaluating the Effect of DA-EPOCH-R Induction Followed by Nivolumab Consolidation in Patients With Newly Diagnosed High Grade B Cell Lymphoma (HGBL) With MYC and BCL2 and/or BCL6 Rearrangements
Brief Title: DA-EPOCH-R Induction Followed by Nivolumab Consolidation in Newly Diagnosed MYC, BCL2 and/or BCL6 Rearranged HGBL
Acronym: HO152
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO152; 2017-003631-12 (EudraCT Number)
Record Dates: First submitted 2018-07-26; First posted 2018-08-08 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Non Hodgkin Lymphoma; Lymphoma, B-Cell; High-grade B-cell Lymphoma; MYC Translocation; BCL-2 Translocation
Keywords: DLBCL; HGBL; BCL-2; BCL-6; double-hit; triple-hit; R-CHOP; DA-EPOCH-R; Nivolumab; PD1/PDL1 expression
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: The trial is designed as a prospective, multicenter, non-randomized phase II trial. All eligible patients will be registered during or after first R-CHOP, but before start of DA-EPOCH-R treatment and before start of nivolumab treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DA-EPOCH-R followed by Nivolumab (Experimental): 5 cycles of DA-EPOCH-R protocol induction, followed with one year Nivolumab consolidation for end-of-induction patients who are in complete metabolic response
  Interventions: Drug: DA-EPOCH-R followed by Nivolumab

INTERVENTIONS:
Drug: DA-EPOCH-R followed by Nivolumab — 5 induction cycles of DA-EPOCH-R protocol, for patient with Deauville imaging response criteria proven complete metabolic response followed with one year Nivolumab consolidation therapy
  Other Names: Opdivo

SUMMARY:
The prognosis of patients with "high-grade B cell lymphoma with cellular myelocytomatosis (MYC) and B cell lymphoma 2 (BCL2) and/or B cell lymphoma 6 (BCL6) rearrangements" (double hit (DH)/triple hit (TH)-HGBL) with rituximab-CHOP (R-CHOP) is dismal as compared to patients with diffuse large B cell lymphoma (DLBCL) without MYC, BCL2 and/or BCL6 rearrangements. Currently, there is no other standard first line treatment for these patients. Dose Adjusted - Etoposide Prednisone Vincristine Cyclophosphamide Doxorubicin - Rituximab (DA-EPOCH-R) and nivolumab are both feasible treatments. Nivolumab may induce auto-immune reactions. DA-EPOCH-R may induce more hematological toxicity than R-CHOP. The hypothesis is that addition of nivolumab to DA-EPOCH-R will contribute to increased survival.

DETAILED DESCRIPTION:
The dismal prognosis of DH-DLBCL patients following standard therapy with R-CHOP (overall survival at 2 years 35% for MYC+ vs 61% for MYC- patients) justifies upfront new treatment approaches.

Attempts have been made to improve prognosis of DH-DLBCL patients with intensified chemotherapy schemes like DA-EPOCH-R, standard treatment of Burkitt lymphoma with high dose multi-agent chemotherapy (R-CODOX-M/R-IVAC) and autologous stem cell transplantation. These treatment schedules seem to prolong disease-free survival (DFS), but relapses do often occur and improved OS has not been achieved. The investigators hypothesize to increase the number of patients in complete remission with DA-EPOCH-R to 65% as compared to 50% for R-CHOP. DA-EPOCH-R is a well-known scheme for the treatment of patients with Burkitt Lymphoma, and is one of the treatment arms of the Hemato-Oncologie voor Volwassenen Nederland (HOVON) 127 protocol. For DH-DLBCL patients the investigators expect that it will improve the complete remission (CR) rate and prolong DFS as compared to R-CHOP as has been shown in several retrospective studies. It is also clear from these studies that relapses still occur and that OS is not improved by chemotherapy only.

The investigators expect to induce deeper remission with DA-EPOCH-R providing the opportunity for nivolumab to consolidate complete remission, prolong DFS, or to induce conversion of minimal residual disease (MRD) positivity to MRD negativity.

A new approach underlying this proposal is to enhance anti-tumor immune responses. Malignancies with MYC aberrations were long thought to be independent of immune responses. However, recently it was shown that MYC expressing lymphoma and leukaemia mouse and human cell lines upregulate programmed death-ligand 1 (PDL1) ("don't find me" signal) and CD47 ("don't eat me" signal) expression. Inactivation of MYC enhanced tumour immune responses in vivo in mice. Moreover, a subset of DLBCL does express PDL1.

No correlation with MYC rearrangements or protein expression has been described in these studies; however, these data suggest that tumours with MYC overexpression may be especially vulnerable to treatment with immune check point inhibitors, providing the rationale for treatment with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for DA-EPOCH-R induction:

* High-grade B-cell lymphoma, with MYC in combination with BCL2 and/or BCL6 rearrangements as assessed by fluorescence in situ hybridization (FISH) according to the WHO 2016 classification including high-grade B-cell lymphoma with MYC and BCL2 rearrangements, transformed from previously untreated FL.
* Age ≥ 18 year.
* Patient started with or has received one course of full dose R-CHOP. [Reversed R-CHOP (cyclophosphamide, vincristine and doxorubicin on day 5) is allowed; local radiation or short course (max 7 days) of steroids (max 100 mg/day) before R-CHOP is allowed. Mini-R-CHOP is not allowed].
* World Health Organization (WHO) performance status 0-3 during or after the first R-CHOP cycle.
* Ann Arbor stage II-IV at diagnosis.
* 18F-FDG PET scan and contrast enhanced CT-scan performed within 21 days before start first cycle of R-CHOP.
* Measurable disease: on contrast enhanced CT-scan at least 1 lesion/node with a long axis of >1.5 cm and at least one 18F-FDG avid lesion.
* Negative pregnancy test at study entry.
* Patient is willing and able to use adequate contraception until 6 months post last treatment administration.
* Written informed consent.
* Patient is capable of giving informed consent.

Inclusion criteria for Nivolumab consolidation:

* Complete metabolic response on end of induction 18F-FDG PET-CT assessed with the Deauville response criteria
* Patient has completed at least R-CHOP plus four cycles of DA-EPOCH-R induction treatment

Exclusion Criteria:

Exclusion Criteria for DA-EPOCH-R induction:

* All histopathological diagnoses other than DH/TH-HGBL (like testicular large B-cell lymphoma or primary mediastinal B-cell lymphoma) according to WHO 2016 classification.
* Known history of indolent lymphoma previously treated with immunochemotherapy.
* Inadequate renal function or creatinine clearance < 30 mL/min (after rehydration). Creatinine clearance (CrCl) may be calculated by Cockcroft -Gault formula: CrCl = (140 - age [in years]) x weight [kg] (x 0.85 for females) (0.815 x serum creatinine [μmol/L])
* Inadequate hepatic function: bilirubin > 3 times upper limit of normal (ULN) (total) except patients with Gilbert's syndrome as defined by > 80% unconjugated bilirubin.
* Inadequate hematological function: absolute neutrophil count (ANC) < 1.0x109/L or platelets < 75x109 /L before R-CHOP unless lymphoma related.
* Central nervous system (CNS) localization of the lymphoma. Cerebrospinal fluid (CSF) analysis before start of treatment is only necessary in case of suspicion of CNS localization.
* Female subject pregnant or breast-feeding.
* History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or stage 0 cervical carcinoma.
* Active symptomatic ischemic heart disease, myocardial infarction, or congestive heart failure within the past year. In case of cardiac history, an echo or multigated acquisition (MUGA) should be obtained and left ventricular ejection fraction (LVEF) should exceed 40% to be eligible.
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, cancer, etc.) that would jeopardize the patient's ability to receive the regimen with reasonable safety.
* HIV positivity.
* Active Hepatitis B or C infection as defined by positive serology and transaminitis. Non-active Hepatitis B carriers may be included if protected
* Severe pulmonary dysfunction (CTCAE grade III-IV).
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior treatment with an anti-PD1, anti-PDL1, anti-PDL2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Severe neurological or psychiatric disease.
* Current participation in another clinical trial interfering with this trial.
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Claustrophobia precluding PET-CT.

Exclusion criteria for Nivolumab consolidation:

* Inadequate renal function or creatinine clearance < 30 mL/min (after rehydration). Creatinine clearance may be calculated by Cockcroft -Gault formula: CrCl = (140 - age [in years]) x weight [kg] (x 0.85 for females) (0.815 x serum creatinine [μmol/L])
* Inadequate hepatic function: bilirubin > 3 times ULN (total) except patients with Gilbert's syndrome as defined by > 80% unconjugated bilirubin.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
12 months DFS from Nivolumab consolidation registration | 12 months
  12 months DFS (defined as time from registration for consolidation to disease relapse or death, whichever comes first) of patients in CMR as assessed by end of DA-EPOCH-R treatment 18F-Fludeoxyglucose Positron Emission Tomography- Computed Tomography (18F-FDG PET-CT)

SECONDARY OUTCOMES:
Complete metabolic response (CMR) rate on 18F-FDG PET-CT after DA-EPOCH-R | at 18 weeks
  CMR rate on 18F-FDG PET-CT after DA-EPOCH-R
18 months Progression-Free Survival (PFS) | 18 months
  18 months PFS (defined as time from registration to disease progression, relapse or death, whichever comes first)
18 months OS | 18 months
  18 months OS (defined as time from registration until death from any cause; patients still alive or lost to follow up are censored at the date they were last known to be alive) of all patients
12 months OSc | 12 months
  12 months overall survival under consolidation (OSc), defined as time from registration for consolidation until death from any cause. Patients still alive or lost to follow up are censored at the date they were last known to be alive
Rate of CTCAE grade >=2 toxicities | During 70 weeks treatment + 100 additional days during follow up
  Rate of CTCAE grade >=2 toxicities
consolidation MRD conversion | 12 months
  Rate of conversion to MRD negativity during consolidation
predictive value of mid-treatment 18F-FDG PET-CT | 2 months
  Assessment of the predictive value of mid-treatment 18F-FDG PET-CT with respect to CMR at the end of DA-EPOCH-R therapy

CONTACTS AND LOCATIONS:
Overall Officials: M. ED Chamuleau, MD PhD, Principal Investigator — VUmc / HOVON
Locations (24):
- Belgium (2):
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Leuven-UZLEUVEN, Leuven
- Netherlands (22):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Almere-FLEVOZIEKENHUIS, Almere Stad
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Goes-ADRZ, Goes
  - NL-Groningen-UMCG, Groningen
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Hoorn-DIJKLANDERHOORN, Hoorn
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Rotterdam-MAASSTADZIEKENHUIS, Rotterdam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Den Haag-HAGA, The Hague
  - NL-Tilburg-ETZ, Tilburg
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle

REFERENCES:
- See also: Website of the HOVON organisation — http://www.hovon.nl